CLINICAL TRIAL: NCT05586542
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter Clinical Study to Assess the Safety of DERMASEAL Advanced Wound Care Dressing for the Treatment of Chronic Non-healing, Neuropathic Diabetic Foot Ulcers
Brief Title: Study to Assess the Safety of DERMASEAL for Diabetic Foot Ulcers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vitruvian Medical Devices, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: VMD2022-001
Record Dates: First submitted 2022-10-16; First posted 2022-10-19 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Foot Ulcer, Diabetic
Keywords: diabetes; non-healing; chronic; skin substitute
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Bronchiolitis Obliterans Syndrome | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: At each site, at least 1 staff member will be identified as the Unblinded Investigational Product Administrator. This site staff member will be responsible for all IP application and wound dressing and undressing at each study visit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard of Care (SOC) (Active Comparator): 1. Wash and sharps debride the target diabetic foot ulcer to remove all non-viable tissue, callus, epibole at wound edges, slough, and debris (at the physician's discretion). The wound margins should be excised to healthy bleeding tissue.
  2. Wash the wound once more with saline to remove remaining debris and confirm hemostasis is achieved, as needed.
  3. Measure wound after debridement.
  4. Place soft silicone contact layer dressing to cover over the wound, secured with adhesive strips.
  5. Cover the contact layer with a hydroconductive wound dressing secured with kerlix gauze and adhesive tape.
  6. Apply the Foot Defender® boot.
  Interventions: Other: Standard of Care
- Plasma Film (Experimental): 1. Wash and sharps debride the target diabetic foot ulcer to remove all non-viable tissue, callus, epibole at wound edges, slough, and debris (at the physician's discretion). The wound margins should be excised to healthy bleeding tissue.
  2. Wash the wound once more with saline to remove remaining debris and confirm hemostasis is achieved, as needed.
  3. Measure wound after debridement.
  4. Place an appropriately sized piece of Plasma Film onto the wound bed. The test agent should be cut to fit the interior of the wound with minimal overlap onto healthy skin.
  5. Place soft silicone contact layer dressing to cover over the wound, secured with adhesive strips.
  6. Cover the contact layer with a hydroconductive wound dressing secured with kerlix gauze and adhesive tape.
  7. Apply the Foot Defender® boot.
  Interventions: Biological: Plasma Film; Other: Standard of Care
- DERMASEAL (Experimental): 1. Wash and sharps debride the target diabetic foot ulcer to remove all non-viable tissue, callus, epibole at wound edges, slough, and debris (at the physician's discretion). The wound margins should be excised to healthy bleeding tissue.
  2. Wash the wound once more with saline to remove remaining debris and confirm hemostasis is achieved, as needed.
  3. Measure wound after debridement.
  4. Place an appropriately sized piece of DERMASEAL onto the wound bed. The test agent should be cut to fit the interior of the wound with minimal overlap onto healthy skin.
  5. Place soft silicone contact layer dressing to cover over the wound, secured with adhesive strips.
  6. Cover the contact layer with a hydroconductive wound dressing secured with kerlix gauze and adhesive tape.
  7. Apply the Foot Defender® boot.
  Interventions: Combination Product: DERMASEAL; Other: Standard of Care

INTERVENTIONS:
Combination Product: DERMASEAL — a novel skin substitute formulated as planar, thin film
  Arms: DERMASEAL
Biological: Plasma Film — a planar, thin film made from human plasma
  Arms: Plasma Film
Other: Standard of Care — standard procedures for managing diabetic foot ulcers including debridement of unhealthy tissue and maintenance of a moist wound environment

SUMMARY:
The goal of this clinical trial is to determine the safety of DERMASEAL for the treatment of non-healing, neuropathic diabetic foot ulcers. The main outcome measure is safety. A total of twenty-four (24) participants will be randomized to receive up to four (4) consecutive weeks of treatment with either standard of care (SOC), plasma film + SOC, or plasma film containing silver microparticles (DERMASEAL) + SOC, with a final follow-up visit 12 weeks after the last treatment.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, multi-center, phase 1 study to evaluate the safety of the DERMASEAL advanced wound care dressing in the treatment of non-healing diabetic foot ulcers located distal to the malleolus in subjects with controlled diabetes mellitus and without significantly compromised arterial circulation. Subjects will be randomized in a 1:1:2 ratio to one of 3 treatment groups:

* SOC alone (n=6)
* SOC + plasma film (n=6)
* SOC + DERMASEAL (n=12)

A subject's study duration will be up to a total of 18 weeks from screening to end of study. This includes a two-week active run-in followed by up to 4 weeks of treatment, plus a final follow-up visit 12 weeks after the last treatment.

The primary endpoint is safety of topically applying a plasma film containing metallic silver microparticles plus fibrin in patients with chronic, non-healing neuropathic diabetic foot ulcers. Secondary endpoints to be assessed in each group include:

1. Percent of study wounds healed during the post-treatment weeks 1 through 4,
2. Time to complete wound closure,
3. Percent area reduction during the post-treatment weeks 2, 4, 6 and 16, and
4. Cost of treatment

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 21 years of age.
2. The subject is able and willing to adhere to study procedures and informed consent is obtained.
3. A non-healing ulcer that is diabetic and neuropathic in origin, located on the foot as defined by beginning >50% below the malleoli of the ankle.
4. Target ulcer surface area between 1 - 10 cm2 after debridement with no active infection.
5. Patients with Type 1 or Type 2 diabetes (criteria for the diagnosis of diabetes mellitus per American Diabetes Association.)
6. Additional wounds may be present but not within 2 cm of the target ulcer.
7. Patient has adequate arterial perfusion of the affected extremity as demonstrated by any one of the following within the past 90 days from the time of screening:

   i. Toe pressure (plethysmography) >50 mm/Hg OR ii. Ankle Brachial Index (ABI) with results ≥ 0.70 and ≤ 1.2 OR iii. TcpO2 ≥30 mm Hg from the foot OR iv. Doppler arterial waveforms consistent with adequate flow in the foot (biphasic or triphasic waveforms at the ankle of affected leg)
8. Target ulcer involves a full thickness skin loss, WITHOUT exposure of tendon, muscle, or bone (University of Texas Grade 1-A or Wagner Grade 1) that has been present ≥ 4 weeks. at the time of screening.
9. HbA1c <10% taken within 30 days prior to Visit 3.
10. Serum creatinine <3.0 mg/dl within the last 6 months.
11. Willing and able (subject or responsible caregiver) to maintain required off-loading (as applicable for the location of the ulcer).
12. Negative urine pregnancy test at Visit 3 for women of childbearing potential. i) Women participants are considered of non-childbearing potential if they are pre-menopausal with a documented hysterectomy or bilateral oophorectomy; or post-menopausal defined as the cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; or have a serum Follicle Stimulating Hormone level confirming the post-menopausal state.

Exclusion Criteria:

1. Suspected or confirmed signs/symptoms of wound infection (subjects may be rescreened if the infection has been treated.) Infection is defined as, for example:

   i. purulence, erythema, cellulitis, excessively high temperatures in/around the ulcer, atypical smell, and/or excessive pain in/around the ulcer (infection may be treated and subject reconsidered for study participation).

   ii. osteomyelitis, with necrotic soft bone. (x-ray to be obtained if in the opinion of the investigator additional confirmation of diagnosis required)
2. Patients presenting with an ulcer probing to tendon, capsule or bone (University of Texas Grade 2 or 3 or deep Wagner 2 or 3).
3. Hypersensitivity to silver or fresh frozen plasma.
4. The subject was previously entered into this study or had participated in any study drug or medical device study within 30 days of screening.
5. Currently on a treatment regimen or medications which in the opinion of the investigator are known to interfere with wound healing (for example: cancer chemotherapy or equivalent immunosuppressants, systemic steroids > 10 days of treatment, cytostatic drugs, cyclooxygenase-2 inhibitors, or radiation therapy).
6. Excessive lymphedema that in the opinion of the investigator will interfere with wound healing.
7. A cognitive, physical, or psychological condition interfering with subject's ability to comply with the treatment regimen.
8. Active Charcot foot or unstable Charcot that in the opinion of the investigator will inhibit wound healing.
9. Wounds secondary to vasculitis, neoplasms, or hematological disorders. Patients on anticoagulation medication will as in any surgical procedure, be monitored according to the protocols employed at the enrolling center.
10. An ulcer that in the opinion of the investigator is not associated with the subject's diabetic neuropathic condition.
11. Subjects is on dialysis.
12. History of radiation to the target foot.
13. Patients with uncontrolled autoimmune connective tissue diseases.
14. Patients who are pregnant, breast feeding, or unwilling to practice contraceptive methods during participation in the study, if applicable. Effective methods of contraception include:

    i. oral, injectable, or implanted hormonal contraceptives ii. intrauterine device or system, iii. barrier method with spermicide, or iv. bilateral tubal occlusion.
15. Patients with uncontrolled anemia (Hgb<10 g/dL in women; <12 g/dL in men) at Screening.
16. Severe malnutrition (serum albumin ≤2.0 with a normal C-reactive protein).
17. Wounds healed by >30% in area following the 2-week, active run-in period as measured during Visit 3.
18. Use of hyperbaric oxygen, and active dressings that include growth factors, engineered tissues, or skin substitutes (e.g., Regranex, Dermagraft, Apligraf, etc.) within 30 days of study screening.
19. Wounds >5 mm deep after sharp debridement.
20. Clinical suspicion of skin cancer at or near the ulcer location which has not been ruled out by biopsy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 16 weeks
  Review of adverse events associated with the topical application of a plasma film containing metallic silver microparticles in patients with chronic non-healing neuropathic diabetic foot ulcers.

SECONDARY OUTCOMES:
Wound healing | 4 weeks
  Percent of study wounds healed during the post-treatment weeks 1 through 4.
Complete wound closure | 16 weeks
  Time to complete wound closure.
Wound area change | 16 weeks
  Percent area change during the post-treatment weeks 2, 4, 6 and 16
Cost | 16 weeks
  Total indirect and direct costs of subject treatment during the study period

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Limb Preservation Platform, Inc., Fresno, California
  - Doctors Research Network, South Miami, Florida
  - Lower Extremity Institute for Research and Therapy, LLC, Boardman, Ohio
  - Futuro Clinical Trials, LLC, McAllen, Texas

IPD SHARING:
Plan to Share IPD: No